CLINICAL TRIAL: NCT04672746
Title: The Medical Peer-delivered Intervention of Brief Motivational Interviewing Via Instant Messaging Interaction in Reducing the Drug Abuse Among Youth in Hong Kong: A Randomized Controlled Trial
Brief Title: Peer-delivered Brief Motivational Interviewing Via Instant Messaging Interaction in Reducing the Drug Abuse Among Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MedPAC-RCT
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Drug Abuse; Adolescent Behavior
Keywords: drug abuse; brief motivational interview; peer counselling; instant messaging; adolescent
MeSH Terms: conditions — Substance-Related Disorders; Adolescent Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief MI interaction via instant communication (Experimental): The interaction communication using brief motivational interviewing will be applied via the chatting function of instant messaging apps (e.g., WhatsApp, WeChat). The intervention will last for 6 month with a frequency of at least twice a week.
  Interventions: Behavioral: Brief MI interaction via instant communication
- General health information (Placebo Comparator): The subjects will receive general health information via SMS, such as "do physical exercise for at least 30 min per week will keep you healthy" for 6 month with a frequency of least twice a week.
  Interventions: Behavioral: General health information

INTERVENTIONS:
Behavioral: Brief MI interaction via instant communication — Telephone peer counselling+referral to treatment if required+The interaction communication using brief motivational interviewing via the chatting function of instant messaging apps (e.g., WhatsApp, WeChat). The intervention will last for 6 month with a frequency of at least twice a week.
  Arms: Brief MI interaction via instant communication
Behavioral: General health information — Telephone peer counselling+referral to treatment if required+general health information via SMS, such as "do physical exercise for at least 30 min per week will keep you healthy" for 6 month with a frequency of least twice a week.
  Arms: General health information

SUMMARY:
This is a two-arm, parallel-group, randomized controlled trial with an allocation ratio 1:1, by comparing the 12-month drug abuse reduction between the youth drug abusers who are individually randomized to participate in the intervention group receiving medical peer-delivered intervention of interactive brief motivational interviewing via instant messaging communication and those in the control group receiving general health information.

DETAILED DESCRIPTION:
Introduction Drug abuse is a worldwide problem especially among youth. Due to easy access to a wide range of illicit drugs via multiple approaches in Hong Kong, growing drug abuse is exposing and spreading among the youth. According to the Central Registry of Drug Abuse Report in Hong Kong, 87.3% of drug abusers reported the first abuse of drugs at ages of 25 or below. The comparison of the Central Registry of Drug Abuse between 2014/15 and 2017/18 showed that the number of students claiming to have used drugs has gone up by 23 percent compared to the last survey, and 81% of them started to use drugs at an age younger than 15-year. The early age of first drug use is strongly associated with the risk of developing a substance use disorder in later life. Youth who persistently abuse substances often experience an array of problems, including academic difficulties, health-related problems (including mental health), poor peer relationships, risky sexual behavior, the likelihood of having blood-borne diseases, and involvement with the juvenile justice system. Additionally, there are harmful consequences for family members, the community, and the entire society. The statistics above alarm that youth drug abuse in Hong Kong is becoming a major problem and can not be overlooked.

The combination of medical treatment and counselling is the most common treatment for drug abusers. However, more than half of the youth drug abusers reported never attempting to quit, only 12.2% of youth drug abusers attempted to seek help, and more than 75% did not accept medical treatment as they did not think they were addicted. Although many non-pharmaceutical interventions have been applied, a meta-analysis found that the existing non-pharmaceutical interventions showed insignificant effectiveness in helping youth drug abusers to change their behaviour. One of the major reasons for the failure to assist youth drug abusers to change was that the patient education method may lead the youth abusers resistant to accept the intervention. Previous research has confirmed that the recovery from drug abuse is influenced by the users' intention to change, which is determined directly by their perceptions of anti-drug and their perceived self-efficacy to change. While, drug-abusers' attitudes, social influences, and demographic characteristics have more indirect effects on recovery from drug abuse. Another reason may be that standard interventional content may not be able to meet the personal needs of drug abusers. In addition, the meta-analysis also showed that individual interventions with more than one session had a stronger effect, while previous brief interventions provided insufficient sessions to support the behavior changes among youth abusers. In addition, according to qualitative interviews conducted for youth drug abusers, adolescents were reluctant to seek help from sources that they believed would be judgmental, lacked expertise, personal information exposed or would inform their parents. Given that, more feasible, individualized, and effective non-pharmaceutical interventions should be developed and evaluated to help this youth population to change.

Conceptual framework Medical peer-delivered counselling Comparing with general counselors, the use of peer counselors can increase the appeal of addiction services to youth and young adult users. Since most young people are not eligible to hold positions of power in their society, they find themselves, subject to authority. Such powers differential made communication between adults and youth difficult. When one is trying to engage the youth in drug abuse reduction initiatives, this power differential manifests itself also as a knowledge gap. Comparing with adults, the equality in power status between the youth makes peer-delivered risk communication successful. However, Addiction counseling on drug abuse is more complex compared with smoking cessation or alcohol and requires more professionalism. With the advantages of similar age and capability to better master related knowledge and counseling skills, peers with a medical background can address youths' concerns relevant to their experience.

Instant messaging Given the ubiquity of mobile technology among youth, and the considerable logistical barriers to face-to-face-based care, instant messaging (IM) via mobile applications such as WhatsApp or WeChat is increasingly used as a new strategy for health promotion and to enhance treatment compliance. As reported in the previous study, drug-abusing clients prefer to use online counseling as it was less confronting to traditional forms of counseling by providing a private and emotionally safe environment. Therefore, the interaction via smart phone apps encourages those who are reluctant to get help face-to-face to seek direct anti-drug advice. In addition, another advantage of using instant messaging is to offer quick, real-time interactions, thus delivering continuous professional advice and personalised support to drug abusers to help them overcome withdrawal symptoms.

Brief Motivational Interviewing Motivational interviewing (MI) was originally developed in the field of alcohol abuse and found to be transferable to other health-related behaviors. Differing from prevailing patient education methods, MI is a directive, client-centered counselling strategy that encourages clients to explore and resolve their ambivalence and promotes their confidence in their ability to change their behaviour. Brief MI, with the advantage of manpower saving, shares the same core as MI that individuals are advocates to initiate and continue behavioural change, and yet often in a state of ambivalence with fluctuating motivations before the behavioural change. Brief MI emphasizes adopting shorter and simpler strategies, which include opening strategy, a typical day, the good things and the less good things, providing information, the future and the present, exploring concerns, and helping with decision-making. By using these specific techniques in the dynamic and interactive process, brief MI explore and resolve the ambivalence, develop discrepancies between individuals' core belief and the behaviour of not engaging in desirable health-related lifestyle practice, consequently enhancing the confidence and motivation in the behavioural change.

Incorporating of Medical peer counselling, instant messaging, and brief MI in promoting drug abuse reduction among youth In combination, the medical peer-delivered intervention via instant messaging interaction may be more effective in helping drug-abusing youth to eliminate or reduce the fear of personal information exposure, the unknown to expect from the treatment, and the whole lifestyle change, and worries about withdrawal symptoms. This approach has the potential to increase the help-seeking behavior and intention to quit among youth drug abusers who reluctant to seek help from services requiring real-name registration. By using the brief MI strategies, youth drug abusers can be guided to attempt behaviour change step by step, and subsequently, could abstain from drugs with assistance.

As stated above, the proposed intervention may be feasible and own potentially effective in reducing drug abuse among youth. However, according to our literature search, there is a paucity of studies exploring its effectiveness. Given that, this study aims to conduct a randomized controlled trial to inform the effectiveness of a medical peer-delivered intervention of interactive brief motivational interviewing via instant messaging communication in reducing drug abuse among youth in Hong Kong

ELIGIBILITY:
Inclusion Criteria:

* aged ≤ 25 years;
* report taking drugs within the past 30 days;
* be able to speak Cantonese and read traditional Chinese;
* accept to received counseling use messaging apps (such as WhatsApp, WeChat, and SMS text messenger);
* have verbally consented to join the follow-up intervention

Exclusion Criteria:

* have acute psychosis or other mental problems,
* are undergoing other drug abuse recovery treatment.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in drug consumption at 12 months comparing to that at baseline | 12 month
  The participants' changes in drug consumption between baseline and 12 months follow-up measured using a structured-questionnaire gathering the frequency and categoties of drug consumption in the past 30 days. The more frequencies and the more kinds of drug used indicating the higher consumption of drug abuse.

SECONDARY OUTCOMES:
Changes in drug consumption at 6 month comparing to that at baseline | 6 month
  The participants' changes in drug consumption between baseline and 6 months follow-up using using a structured-questionnaire gathering the frequency and categoties of drug consumption in the past 30 days. The more frequencies and the more kinds of drug used indicating the higher consumption of drug abuse.
30 days self-reported drug abstinence at 6 months | 6 month
  The participants' 30 days self-reported drug abstinence at 6 months follow-up measured using using a structured-questionnaire gathering the frequency and categoties of drug consumption in the past 30 days. The self-reported non-drug consumption indicating drug abstinence.
30 days self-reported drug abstinence at 12 months | 12 month
  The participants' 30 days self-reported drug abstinence at 12 months follow-up measured using using a structured-questionnaire gathering the frequency and categoties of drug consumption in the past 30 days. The self-reported non-drug consumption indicating drug abstinence.
Changes in relapse risk among the quitters at 6 months comparing to that at baseline | 6 month
  The participants' changes in relapse risk between baseline and 6 months follow-up measured using the Stimulant Relapse Risk Scale (Chinese version). The scale consists of 27 items and measures the risk of stimulant reuse in 5 dimensions: anxiety and intention to use drug, emotionality problems, compulsivity for drug use, positive expectancies and lack of control over drug, and lack of negative expectancy for drug use.
Changes in relapse risk among the quitters at 12 months comparing to that at baseline | 12 month
  The participants' changes in relapse risk between baseline and 12 months follow-up measured using the Stimulant Relapse Risk Scale (Chinese version). The scale consists of 27 items and measures the risk of stimulant reuse in 5 dimensions: anxiety and intention to use drug, emotionality problems, compulsivity for drug use, positive expectancies and lack of control over drug, and lack of negative expectancy for drug use.
Changes in the contemplation stages at 6 months comparing to that at baseline | 6 month
  The participants' changes in the contemplation stages between baseline,and 6 months follow-up measured using the Contemplation Ladder Tool. The tool consists of 5 items which include pre-contemplation stage, contemplation stage, decision stage, action stage, and maintenance stage.
Changes in the contemplation stages at 12 months comparing to that at baseline | 12 month
  The participants' changes in the contemplation stages between baseline, and 12 months follow-up measured using the Contemplation Ladder Tool. The tool consists of 5 items which include pre-contemplation stage, contemplation stage, decision stage, action stage, and maintenance stage.
Changes of motivation towards solving the problem at 6 months comparing to that at baseline | 6 month
  Participants' changes of motivation towards solving the problem between baseline and 6 months follow up measured using the Chinese version of Treatment Needs/Motivation Scales (TCU MOTForm). The scale consists of 36 items with 5 dimensions: Problem Recognition (PR), Desire for Help (DH), Treatment Readiness (TR), Pressures for Treatment (PT), and Treatment Needs (TN), which are using a 5-likert score. The score of the scale ranges from 36 to 180, with higher score indicating a higher motivation towards solving the problem.
Changes of motivation towards solving the problem at 12 months comparing to that at baseline | 12 month
  Participants' changes of motivation towards solving the problem between baseline and 12 months follow up measured using the Chinese version of Treatment Needs/Motivation Scales (TCU MOTForm). The scale consists of 36 items with 5 dimensions: Problem Recognition (PR), Desire for Help (DH), Treatment Readiness (TR), Pressures for Treatment (PT), and Treatment Needs (TN), which are using a 5-likert score. The score of the scale ranges from 36 to 180, with higher score indicating a higher motivation towards solving the problem.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Shuk Ting Cheung, PhD, Study Director — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient-level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project is completed and the results of the project have been published.
Access Criteria: Request could be sent to Principal Investigator (william3@hku.hk)